CLINICAL TRIAL: NCT03220230
Title: NON INTERVENTIONAL MULTICENTER STUDY, FOR THE VALIDATION OF MOLECULAR DIAGNOSTIC TECHNOLOGIES IN SUBJECTS WITH NON SMALL CELL LUNG CANCER (NSCLC) PROTOCOL N° X9001083
Brief Title: Validation of Molecular Diagnostic Thecnologies for Lung Cancer Patients.
Acronym: NIRVANA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001083; NIRVANA (Other: Alias Study Number)
Record Dates: First submitted 2017-07-05; First posted 2017-07-18 (Actual); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Lung Neoplasms
Keywords: Next generation sequencing; Lung cancer; target therapies
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tumor tissue whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
This is a non-interventional multi-center with investigational sites in Chile and Brasil diagnostic study to validate novel diagnostic technologies, such as Next Generation Sequencing (NGS) from both tissue and blood compared to the current gold standard. As a non-interventional study, patients will receive the treatment indicated by their doctor independently of their participation on this study.

Many cancer cells look the same under the microscope. But as these cells are studied at the molecular level, some genetic alterations or defects that are more common to certain types of cancer are identified. In some cases, these defects are what make the cells grow and multiply abnormally.

Biomarkers are the molecular fingerprints of these genetic defects. By testing a sample of your tumor for biomarkers, doctors can learn if your cancer has one of these defects, and that may point to a specific treatment choice.

One of the genetic biomarkers that are believed to cause some cancers to grow is the ALK fusion gene. About 3% to 5% of people with NSCLC may test positive for ALK. ROS1 is a receptor found in 1 to 2% of people with this type of cancer.

The present study is designed to advance the molecular testing methodologies to identify ALK+ and ROS1+ NSCLC patients.

A positive correlation with these new technologies will mean an efficient, more accurate diagnostic test, which could impact a greater number of cancer patients around world.

DETAILED DESCRIPTION:
B. Lung Cancer Non-small cell lung cancer (NSCLC) is a common cause of cancer mortality throughout the world. In 2007, there were 1.5 million new lung cancer cases diagnosed worldwide, including around 733,100 cases in the South American Region.6

Approximately 85% of lung cancer is histologically defined as non small cell and the remaining 14% as small cell. The majority of patients with NSCLC present with inoperable locally advanced (Stage IIIB) or metastatic (Stage IV) disease for which no curative treatment is yet available. In newly diagnosed patients with good performance status, platinum based doublet-combination chemotherapies are associated with a median overall survival (OS) of 7.4 to 9.9 months. 7, 8, 9, 10, 11, 12 Therefore, newer agents with novel mechanisms of action are still desperately needed for this serious life-threatening disease. 15,16

The rapid and efficient identification of key driver genes in non-small-cell lung cancer (NSCLC) is becoming increasingly important.17 Clinical screening efforts have revealed that the most common mutations in lung cancer specimens involve EGFR and KRAS, along with 10 other genes that show a prevalence of mutation in 5% or less of tumors. The ALK gene is rearranged in around 3%-5% of patients with NSCLC and has been the focus of intense basic and clinical research, suggesting that the frequency of the gene rearrangement is similar in Asian and Western patients.

ROS1 is a receptor tyrosine kinase of the insulin receptor family. Chromosomal rearrangements involving the ROS1 gene were originally described in glioblastomas, where ROS1 (chromosome 6q22) is fused to the FIG gene (chromosome 6q22 immediately adjacent to ROS1), 16 and have been shown to be transforming in transgenic mice.17 More recently, ROS1 fusions were identified as potential driver mutations in an NSCLC cell line (HCC78; SLC34A2-ROS1) and an NSCLC patient sample (CD74-ROS1). 18 These fusions led to constitutive kinase activity and were associated with sensitivity in vitro and in vivo to crizotinib. As of December 2013, 16 different variants have been found.16, 17, 18

The present study is designed to advance the molecular testing methodologies to identify ALK+ and ROS1+ NSCLC patients. Advanced next generation sequencing screening methodologies will be used to identify NSCLC patients whose tumors contain a ROS1 gene inversion or translocation or an ALK translocation.

A parallel test for ALK+ by either the Abbott ALK FISH test or the Ventana ALK IHC test is necessary to validate the NGS test in all samples. A parallel test for ROS1+ by either the Kreatech FISH test or the D4D6 ROS1 IHC test may be necessary to validate the NGS test in all samples.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 years of age or older.
* Patients with histologically or cytological proven diagnosis of NSCLC, pathologically identified as adenocarcinoma.
* Patient naïve in lung cancer treatment
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the study prior to enrollment.
* Patients must give consent to the research use of their archived or tumor FFPE tissue, and if available, 2 blood tubes.

Exclusion Criteria:

* Prior chemotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 4240 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Ricardo Armisen, MD, PhD, Study Chair — CEMP Pfizer Chile
Locations (37):
- Brazil (19):
  - Centro Regional Integrado de Oncologia, Fortaleza, Caera
  - Instituto Goiano de Oncología e Hematologia, Aparecida de Goiana, Goiás
  - Hospital Luxemburgo, Belo Horizonte, Minas Gerais
  - Hospital Felicio Rocho, Belo Horizonte /MG, Minas Gerais
  - Instituto de Cancer de Londrina, Londrina, Paraná
  - Centro de Pesquisa da Universidade Federal de Sao Paulo - UNIFESP, São Paulo, VILA Clementino
  - Fundaçao Pio XII, Hospital do Cancer de Barretos, Barretos
  - Liga Paranaense de Combate ao Cancer Hospital Erasto Gaetner, Curtiba-PR
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alegre (ISCMPA) - Hospital Santa Rita, Porto Alegre
  - Instituto de Medicina Integral Prof. Fernando Figueira - IMIP, Recife
  - Instituto COI de Pesquisa Educacao e Gestao, Rio de Janeiro
  - Hospital Da Bahia, Salvador
  - Hospital Santa Izabel, Salvador
  - Nucleo de Oncologia da Bahia, Salvador
  - Instituto de Oncologia de Sorocaba - ONCO Clinicas Especializadas SC Ltda, São Paulo
  - A.C. Camargo Cancer Center, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo/SP
- Chile (9):
  - Hospital Base de Puerto Montt, Port Montt, Los Lagos Region
  - Hospital Base de Valdivia, Valdivia, Los Lagos Region
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco, Ranco
  - Centro Internacional de Estudios Clinicos, Santiago, RM
  - Hospital Clinico Universidad de Chile, Seccion de Oncologia, Independencia, Santiago, RM
  - Hospital Base de Arica, Arica
  - Hosp Regional de Concepcion, Concepción
  - Universidad Católica del Norte, Coquimbo
  - Instituto Nacional Del Torax, Santiago
- Peru (9):
  - Hospital Carlos Alberto Seguin Escobedo, Arequipa
  - Hospital Nacional Hipolito Unanue, El Agustino
  - Clinica San Felipe, Lima
  - Hospital Central de la Fuerza Aerea Peruana, Lima
  - Instituto Nacional de Enfermedales Neoplasicas (INEN), Lima
  - Oncosalud, Lima
  - Unidad de Investigacion de la Clinica Internacional - Sede San Borja, Lima
  - Clínica Quirurgica Santa Maria, Lima
  - Centro de Investigación Clínica Trujillo E.I.R.L., Trujillo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001083

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Small Cell Lung Cancer Participants: Tissue and blood samples of participants with non-small cell lung cancer (NSCLC) were collected and analyzed to validate new molecular diagnostic technologies (such as Next Generation Sequencing [NGS]) and to compare their performance with the available standard tests. Participants were not treated or affected and only participated in the study for the initial samples and clinical parameters collection.
Period: Overall Study
Arm/Group | Non-Small Cell Lung Cancer Participants
Started | 4240
Completed | 4240
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all NSCLC participants who satisfied all inclusion and exclusion criteria.
Groups:
- Non-Small Cell Lung Cancer Participants: Tissue and blood samples of participants with NSCLC were collected and analyzed to validate new molecular diagnostic technologies (such as NGS) and to compare their performance with the available standard tests. Participants were not treated or affected and only participated in the study for the initial samples and clinical parameters collection.
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 4240
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.998 (11.495)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2011
  Male | 2229
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 27
  Black | 68
  Caucasian | 511
  More than one race | 3236
  Native Indian | 10
  Other | 388

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prevalence of Anaplastic Lymphoma Kinase (ALK) Biomarker
Description: ALK status was measured by NGS- Oncomine focus assay (OFA) and Immuno histo chemistry (IHC) Ventana. Ventana -ALK and NGS-OFA were the assay procedures performed for ALK. The corresponding analysis of a specimen had 2 possible test results including ALK positive and ALK negative. True positives (tp) were defined as NGS-OFA and Ventana positive results, whereas false negatives (fn) were defined as NGS-OFA negative results and IHC-Ventana positive results. False positives (fp) were defined as NGS-OFA positive results and IHC-Ventana negative results. True negatives (tn) were defined as NGS-OFA and IHC Ventana negative results.
Time Frame: 40 months
Population: Per protocol analysis set included all participants with valid IHC-Ventana and NGS-OFA results.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 1450
Participants
  ALK-true positive | 45
  ALK-true negative | 1346
  ALK-false positives | 21
  ALK-false negative | 38

2. Primary Outcome: Percentage of Concordance (Agreement) Between Ventana and NGS ALK Result
Description: In this outcome measure, index of concordance with accuracy, sensitivity, specificity, positive predictive value and negative predictive value were measured. Accuracy (Acc): [tp+tn]/[tp+fp+fn+tn] *100; Sensitivity (Ss): tp/[tp+fn] *100; Specificity (Sp): tn/[fp+tn] *100; Positive Predictive Value (PPV): tp/[tp+fp] *100; Negative Predictive Value (NPV): tn/[fn+tn] *100.
Time Frame: 40 months
Population: Per protocol analysis set included all participants with valid IHC-Ventana and NGS-OFA results. Here, "Number analyzed" signifies the number of participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of concordance
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 1450
percentage of concordance
  Accuracy | 95.931 [94.78 to 96.84]
  Sensitivity: number analyzed (Participants) | 83
  Sensitivity | 54.217 [43.548 to 64.512]
  Specificity: number analyzed (Participants) | 1367
  Specificity | 98.464 [97.649 to 99.007]
  Positive Predictive Value: number analyzed (Participants) | 66
  Positive Predictive Value | 68.182 [56.17 to 78.194]
  Negative Predictive Value: number analyzed (Participants) | 1384
  Negative Predictive Value | 97.254 [96.244 to 98.003]

3. Secondary Outcome: Number of Participants With Prevalence of Anaplastic Lymphoma Kinase (ALK) Biomarker by Type of Participants
Description: Participants were categorized on the basis of prospective and retrospective. Prospective participants were those participants whose samples were taken after the informed consent. Retrospective participants were those participants whose samples were taken before the date of signature of the informed consent.
Time Frame: 40 months
Population: Per protocol analysis set included all participants with valid IHC-Ventana and NGS-OFA results. Here, "Overall Number of Participants Analyzed" participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 83
Participants
  Retrospective | 49
  Prospective | 34

4. Secondary Outcome: Number of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Smoking (Tobacco Use) History
Description: The categories of smoker (tobacco use) were as follows: Never Smoker: No smoking exposure, Current Smoker: Currently uses tobacco in either cigarette, cigar or similar method (tobacco chewers excluded), Former Smoker: Participant at one time smoked but then later quit. Smoking status unknown: Participant whose smoking status is unknown.
Time Frame: 40 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 83
Participants
  Tobacco Use: Current | 9
  Tobacco Use: Former | 32
  Tobacco Use: Never | 31
  Tobacco Use: None | 11

5. Secondary Outcome: Number of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Stage and Classification of Biopsy
Description: Stage was defined at time of initial diagnosis of NSCLC and participants were staged according to the guidelines set by the NCCN version 7.2015. Participant's stage was categorized as: stage 0, stage IA, stage IB, stage IIA, stage IIB, stage IIIA, stage IIIB, and stage IV. Biopsy NSCLC class was categorized as adenocarcinoma, neuroendocrine tumors, other known type of NSCLC and squamous cell carcinoma.
Time Frame: 40 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 83
Participants
  Biopsy Stage: IA | 2
  Biopsy Stage: IB | 3
  Biopsy Stage: IIA | 1
  Biopsy Stage: IIB | 1
  Biopsy Stage: IIIA | 7
  Biopsy Stage: IIIB | 7
  Biopsy Stage: IV | 52
  Biopsy Stage: None | 10
  Biopsy NSCLC class: adenocarcinoma | 74
  Biopsy NSCLC class: neuroendocrine tumors | 1
  Biopsy NSCLC class: other known type of NSCLC | 2
  Biopsy NSCLC class: squamous cell carcinoma | 6

6. Secondary Outcome: Number of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Location
Description: Locations were categorized as lungs, pleura, node mediastinal and others.
Time Frame: 40 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 83
Participants
  Lungs | 56
  Pleura | 11
  Other | 9
  Node Mediastinal | 7

7. Secondary Outcome: Number of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Gender and Age
Description: In this outcome measure, participants were categorized according to their gender (female/male) and different age ranges (18-30 / 31-40 / 41-60 / 60 and above).
Time Frame: 40 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 83
Participants
  Gender: Male | 28
  Gender: Female | 55
  Age range: 18-30 years | 1
  Age range: 31-40 years | 7
  Age range: 41-60 years | 37
  Age range: Above 61 years | 38

ADVERSE EVENTS:
Time Frame: Up to 40 months
Arm/Group | Non-Small Cell Lung Cancer Participants
All-Cause Mortality (participants affected / at risk) | 0/4240
Serious Adverse Events (participants affected / at risk) | 0/4240
Other Adverse Events (participants affected / at risk) | 0/4240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03220230/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03220230/SAP_001.pdf